CLINICAL TRIAL: NCT04665635
Title: Comparison of Rectosigmoid Resection and Seromuscular Tumor Shaving Methods in Ovarian Cancer Surgery (BROSEOC)
Brief Title: Rectosigmoid Resection vs Seromuscular Tumor Shaving in Ovarian Cancer Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Ghanim Khatib, Associate professor, MD, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 105/17- Ov01
Record Dates: First submitted 2020-11-30; First posted 2020-12-11 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Epithelial Ovarian Cancer; Rectosigmoid Cancer Metastatic
Keywords: epithelial ovarian cancer; Rectosigmoid resection; Seromuscular tumor shaving; recurrence
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rectosigmoid resection (Active Comparator)
  Interventions: Procedure: Rectosigmoid resection
- Rectosigmoid seromuscular tumor shaving (Active Comparator)
  Interventions: Procedure: Rectosigmoid resection

INTERVENTIONS:
Procedure: Rectosigmoid resection — Most of the colorectal involvements are observed in the seromuscular layer. In seromuscular infiltration, resection of the rectosigmoid colon or shaving of tumoral implants without resection can be performed.
  Other Names: Rectosigmoid seromuscular tumor shaving

SUMMARY:
Ovarian cancer is the most common cause of death in gynecological cancer. Approximately 75% of epithelial ovarian cancers are detected at an advanced stage. Metastasis and spread are mostly through transperitoneal planting and neighborhood by shedding from the ovarian surface. Metastasis mostly occurs in the peritoneum, omentum, and intestines. The rectosigmoid colon is the main part of the intestine affected by metastasis due to its neighborhood.

Treatment in ovarian cancer consists of a combination of cytoreduction surgery and platinum-based chemotherapy. Surgery is the basis of the treatment, and the main goal is to achieve no residual visible tumor (complete cytoreduction: R0). The residual tumor is one of the main factors affecting survival and reflects the possibilities of the surgical center and the team. Multiple surgical procedures (total hysterectomy, bilateral salpingo-oophorectomy, total omentectomy, peritonectomy, retroperitoneal lymphadenectomies such as pelvic and paraaortic, bowel resections, splenectomy, distal pancreatectomy, various resections related to the bladder, liver, stomach, and diaphragm) may be required to achieve complete or optimal cytoreduction.

In the involvement of the rectosigmoid colon, primarily the serosa, then the muscular layer and finally the mucosa are infiltrated due to the nature of the spread, and therefore most of the involvement is observed in the seromuscular layer. In seromuscular infiltration, resection of the rectosigmoid colon or shaving of tumoral implants without resection can be performed. There are advantages and disadvantages of each method in terms of morbidity. Although there are retrospective studies evaluating recurrence and survival between both methods, as far as investigators know, no randomized prospective studies have been conducted comparing these two methods. The investigators designed this study to compare these two methods successfully applied in our clinic in a prospective randomized study.

ELIGIBILITY:
Inclusion Criteria:

* Epithelial ovarian cancer
* Negative colonoscopy ( no mucosal involvement)
* Intraoperative confirmed serosal or seromuscular rectosigmoid infiltration
* ECOG <3
* ASA <3

Exclusion Criteria:

* Nonepithelial ovarian cancers
* Rectosigmoid mucosal infiltration
* Total or subtotal colectomy necessitating large bowel infiltrations
* ECOG >2
* ASA >2

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Local pelvic recurrence | 0-60 months.
  Only the pelvic recurrences determined after the last chemotherapy cycle.
Recurrence-free survival | 0-60 months.
  The time from the last chemotherapy cycle to determination of any recurrence in any location.

SECONDARY OUTCOMES:
Cancer specific survival | 0-100 months
  Time from diagnosis to the death date due to ovarian cancer.
Surgery related morbidities | 90 days.
  Any surgery related morbidity during 90 days.
Health related Quality of life | 0-24 months.
  HRQoL will be assessed with the European Organization for Research and Treatment of Cancer (EORTC) core questionnaire (EORTC QLQ-C30 version 3.0).The QLQ-C30 is a 30-item questionnaire that includes five multiitem functional scales (physical, role, cognitive, emotional, and social), three multi-item symptom scales (fatigue, nausea and vomiting, and pain), five single-item symptom scales (dyspnoea, insomnia, appetite loss, constipation, and diarrhoea), a question on financial impact; and a two-item global quality of life scale.The questionnaire generally has a four-point response scale (1 = "not at all", 4 = "very much").The questionnaire is planned to be performed within 1-2 weeks prior to the surgery (baseline), after 3-4 weeks of surgery before starting of adjuvant chemotherapy, at the end of adjuvant chemotherapy, and every three months in follow-up, until two years of follow-up.
Overall survival | 0-100 months.
  Time from diagnosis to the death date due to any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Cukurova University, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Background] Erkilinc S, Karatasli V, Demir B, Cakir I, Can B, Karadeniz T, Gokcu M, Sanci M. Rectosigmoidectomy and Douglas Peritonectomy in the Management of Serosal Implants in Advanced-Stage Ovarian Cancer Surgery: Survival and Surgical Outcomes. Int J Gynecol Cancer. 2018 Nov;28(9):1699-1705. doi: 10.1097/IGC.0000000000001368. PMID 30371561
- [Result] Gallotta V, Fanfani F, Vizzielli G, Panico G, Rossitto C, Gagliardi ML, Margariti PA, Salerno MG, Zannoni GF, Pacelli F, Scambia G, Fagotti A. Douglas peritonectomy compared to recto-sigmoid resection in optimally cytoreduced advanced ovarian cancer patients: analysis of morbidity and oncological outcome. Eur J Surg Oncol. 2011 Dec;37(12):1085-92. doi: 10.1016/j.ejso.2011.09.003. Epub 2011 Sep 25. PMID 21945640
- [Result] Aletti GD, Podratz KC, Jones MB, Cliby WA. Role of rectosigmoidectomy and stripping of pelvic peritoneum in outcomes of patients with advanced ovarian cancer. J Am Coll Surg. 2006 Oct;203(4):521-6. doi: 10.1016/j.jamcollsurg.2006.06.027. Epub 2006 Aug 23. PMID 17000396